CLINICAL TRIAL: NCT04663165
Title: Biomarkers in Gingival Exudate and Blood Serum Before and After Surgical Treatment of Periodontitis
Brief Title: Biomarkers for Periodontitis Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Holmlund (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Anders Holmlund, Primary Investigator, Associated Professor, Region Gävleborg
Organization: Region Gävleborg (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 476871q
Record Dates: First submitted 2020-11-12; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Periodontitis
Keywords: Periodontitis; Gingival crevicular fluid (GCF); Serum; Inflammation
MeSH Terms: conditions — Periodontitis; Inflammation

STUDY DESIGN:
Intervention Model Description: a clinical prospective interventional study with longterm follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flap surgery alone (Other): Access flap
  Interventions: Procedure: Periodontal surgery
- Flap surgery with adjunctive EMD (Other): Access flap and adjunctive enamel matrix derivative
  Interventions: Procedure: Regenerative periodontal surgery

INTERVENTIONS:
Procedure: Periodontal surgery — Flap surgery at teeth with periodontal pocket depth 5 mm or more with additional bleeding or pus on probing. Elimination of dental calculus and granulation tissue as well as scaling of the root surface with scalers and ultrasonic device. Flap closure with non-resorbable sutures.
  Arms: Flap surgery alone
Procedure: Regenerative periodontal surgery — Flap surgery at teeth with periodontal pocket depth 5 mm or more with additional bleeding or pus on probing combined with vertical bone defect of 4mm or more. After elimination of dental calculus and granulation tissue as well as scaling of the root surface with scalers and ultrasonic device, adjunctive treatment with EDTA gel applied to root surface for two minutes, followed by rinsing with saline solution. Finally, application of enamel matrix derivative on a blood free root surface, followed by flap closure with non-resorbable sutures.
  Arms: Flap surgery with adjunctive EMD

SUMMARY:
In this clinical study, we have collected GCF at diseased teeth and at the same time drawn blood, both before and at 3, 6 and 12 months after periodontal surgical treatment. This give us the opportunity to investigate if periodontal treatment could reduce inflammatory biomarkers in the systemic circulation and if there is a co-variation between biomarkers in GCF and blood.

In part I of this study, we focus on biomarkers from blood serum in patients with periodontitis, before surgical therapy and under a healing period 12 months.

In part II, biomarkers in the locally collected GCF will be analyzed together with clinically reported measurements and compared with biomarkers in blood serum.

Hypothesis are

* Periodontal treatment followed by clinical healing and periodontal health will be associated a change/ reduction in biomarkers in GCF.
* The systemic levels of inflammatory biomarkers may show a delayed response to clinical healing. Periodontal surgical therapy may reduce circulating inflammatory biomarkers that could affect the low-grade chronic inflammation.
* There is a co-variation between inflammatory biomarkers in GCF and the systemic circulation.

DETAILED DESCRIPTION:
Periodontitis, a disease affecting the tissue supporting the tooth, is initiated by microbes colonizing the tooth causing an inflammation of the soft tissue around the tooth. In some sensitive individuals the inflammatory response leads to loss of jawbone, which affect the bone support of the tooth and may end up in loss of teeth. Periodontitis is the sixth most prevalent disease in the world, 40% of the population with affected jawbone support and approximately 10% of the population suffer from severe loss of the supporting jawbone at teeth. Periodontitis may be halted or resolved by removing the microbial biofilm from the teeth root and in severe cases combined with surgical treatment removing inflammatory tissue. The genetic factors explain approximately 50% of the disease, and but the etiology is in parts unclear and effective therapy in sensitive individuals is still missing.

The inflammatory response initiated by microbes leads to degradation of the tooth supporting tissues. The current view is that pro-inflammatory cytokines and prostaglandins, produced by leukocytes and cells of mesenchymal origin in the inflamed tissue are responsible for recruiting and activation of bone-resorbing cells, osteoclasts. The inflammatory biomarkers and tissue degradation products will leak out into the exudate in the gingival pocket next to the root surface. The bone resorption activity connected to changes in biomarkers levels and clinical parameters, during healing after periodontal treatment seem to be of value to study. The analysis of the local exudate (gingival crevicular fluid, GCF) could be used for predicting and monitoring periodontitis, as well as finding new targets for treatment.

Periodontitis could also have a systemic effect, as locally released inflammatory mediators might enter the systemic circulation and influence the development of inflammatory conditions such as cardiovascular disease (CVD), diabetes and rheumatoid arthritis. Earlier studies have shown that a low-grade chronic inflammation plays an important role in the pathogenies in atherosclerosis. Substances that indicate low-grade chronic inflammation in blood serum is for example levels of C-reactive protein (CRP), fibrinogen, and adhesion-molecules, and these biomarkers are related to CVD. The question is if periodontal treatment could change/reduce the systemic inflammatory burden of inflammatory biomarkers (CRP, fibrinogen, interleukins, and matrix metalloproteinases (MMP)).

We know today that there is association between oral health and CVD, but we do not know if the relationship it is of a causal nature. There are some intervention studies that indicate that the oral inflammatory burden may have a systemic effect. To better understand the role of the oral inflammation in development of atherosclerosis, it is important to study biomarkers at different timepoints both from the local sites (GCF) and the general systemic environment in blood. If there is a co-variation in levels of inflammatory biomarkers locally in the GCF and in the systemic circulation, this could be a strong indication of a more causal nature of the association, but we need more studies.

The value of the study is to better understand what drives the local disease progression in periodontitis and also increase the knowledge by which mechanism the oral inflammation could exert its systemic effect. Measuring levels of biomarkers in GCF and serum at several timepoints after treatment we may contribute with new insights in the role of inflammatory inducing molecules in periodontal disease, but also if there exists any systemic effect from locally released inflammatory mediators. The possibility that some molecules co-variate with disease progression or regression is of great value.

The possible co-variation of molecules with disease progression or regression is important knowledge in understanding how oral infection may affect the general health.

Part I: Serum biomarkers for periodontitis relapse Part II: GCF biomarkers for periodontal healing and relapse

This is a prospective clinical intervention study to investigate healing of severe periodontitis sites after periodontal surgical therapy and in what extent the clinical healing is associated with changes of the inflammatory expression of biomarkers in gingival crevicular fluid (GCF) and in blood serum.

21 patients were recruited consecutively and treated surgically of one experienced specialist in periodontology. Two teeth in different quadrants per patient, with the deepest pocket measured, were selected and included in the study. Periodontal surgery was performed and at 13 of the teeth an additional treatment with enamel matrix derivative (EMD/Emdogain®) were performed. Registration of full mouth plaque score (FMPS), periodontal pocket depth (PPD), bleeding on probing (BOP) or pus were performed before surgery, after 3, 6 and 12 months. Radiographs were taken at examination before treatment and at the follow-up at 12 months.

Blood samples and samples of gingival crevicular fluid (GCF) were collected before and at the follow-up visits 3, 6 and 12 months after surgical treatment. GCF samples was labelled and stored at -80°C.

Blood samples were drawn and handled by the chemical laboratory at Gävle hospital in conjunction to therapy and follow-up points. Blood were collected from each patient and 5x1mL serum was labelled and stored at -80°C.

Protein analysis on blood sera and GCF performed and concentrations of 92 proteins were assessed by proximity extension assay (Olink Bioscience, Sweden) using the Inflammation panel.

Vascular Injury Panel 2 Human Kit (Meso Scale Diagnostics) were used to assess concentration of C-Reactive Protein (CRP), Intercellular Adhesion Molecule-1 (ICAM-1), Serum Amyloid A (SAA) and Vascular Cell Adhesion Molecule-1 (VCAM-1) in sera.

ELIGIBILITY:
Inclusion Criteria:

* patient with diagnosed periodontitis
* at least three teeth with ≥ 4mm loss of bone support detected at radiograph, combined with periodontal pocket depth ≥5mm and bleeding on probing and/or pus, in two quadrants

Exclusion Criteria:

* periodontal therapy the last 3 months
* intake of antibiotic the last 3 months
* intake of anti-inflammatory drug the last 2 weeks before collection of samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02-04 (Actual); Primary Completion 2013-09-23 (Actual); Study Completion 2015-01-12 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) 3 months | between baseline and 3 months after treatment
  Change in BOP
Bleeding on probing (BOP) 6 months | between baseline and 6 months after treatment
  Change in BOP
Bleeding on probing (BOP) 12 months | between baseline and 12 months after treatment
  Change in BOP
Periodontal pocket depth (PPD) 3 months | between baseline and 3 months after treatment
  Change in PPD
Periodontal pocket depth (PPD) 6 months | between baseline and 6 months after treatment
  Change in PPD
Periodontal pocket depth (PPD) 12 months | between baseline and 12 months after treatment
  Change in PPD
Plaque Index (PLI) 3 months | between baseline and 3 months after treatment
  Change in PLI
Plaque Index (PLI) 6 months | between baseline and 6 months after treatment
  Change in PLI
Plaque Index (PLI) 12 months | between baseline and 12 months after treatment
  Change in PLI
Biomarkers in blood serum 3 months | between baseline and 3 months after treatment
  Change in serum protein profile using Inflammation panel (92 proteins) by Olink Bioscience plus V-PLEX Vascular Injury Panel 2 Human Kit to assess concentration of CRP, ICAM-1, SAA and VCAM-1.
Biomarkers in blood serum 6 months | between baseline and 6 months after treatment
  Change in serum protein profile using Inflammation panel (92 proteins) by Olink Bioscience plus V-PLEX Vascular Injury Panel 2 Human Kit to assess concentration of CRP, ICAM-1, SAA and VCAM-1.
Biomarkers in blood serum 12 months | between baseline and 12 months after treatment
  Change in serum protein profile using Inflammation panel (92 proteins) by Olink Bioscience plus V-PLEX Vascular Injury Panel 2 Human Kit to assess concentration of CRP, ICAM-1, SAA and VCAM-1.
Biomarkers in gingival crevicular fluid (GCF) 3 months | between baseline and 3 months after treatment
  Change in GCF protein profile using Inflammation panel (92 proteins) by Olink Bioscience.
Biomarkers in gingival crevicular fluid (GCF) 6 months | between baseline and 6 months after treatment
  Change in GCF protein profile using Inflammation panel (92 proteins) by Olink Bioscience.
Biomarkers in gingival crevicular fluid (GCF) 12 months | between baseline and 12 months after treatment
  Change in GCF protein profile using Inflammation panel (92 proteins) by Olink Bioscience.

SECONDARY OUTCOMES:
Association between BOP and serum protein profile 3 months | between baseline and 3 months after treatment
  Change in serum protein profile in relation to the clinical parameter bleeding on probing (BOP)
Association between BOP and serum protein profile 6 months | between baseline and 6 months after treatment
  Change in serum protein profile in relation to the clinical parameter bleeding on probing (BOP)
Association between BOP and serum protein profile 12 months | between baseline and 12 months after treatment
  Change in serum protein profile in relation to the clinical parameter bleeding on probing (BOP)
Association between PPD and serum protein profile 3 months | between baseline and 3 months after treatment
  Change in serum protein profile in relation to the clinical parameter periodontal pocket depth (PPD)
Association between PPD and serum protein profile 6 months | between baseline and 6 months after treatment
  Change in serum protein profile in relation to the clinical parameter periodontal pocket depth (PPD)
Association between PPD and serum protein profile 12 months | between baseline and 12 months after treatment
  Change in serum protein profile in relation to the clinical parameter periodontal pocket depth (PPD)
Association between BOP and GCF protein profile 3 months | between baseline and 3 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters bleeding on probing (BOP)
Association between BOP and GCF protein profile 6 months | between baseline and 6 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters bleeding on probing (BOP)
Association between BOP and GCF protein profile 12 months | between baseline and 12 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters bleeding on probing (BOP)
Association between PPD and GCF protein profile 3 months | between baseline and 3 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters probing pocket depth (PPD)
Association between PPD and GCF protein profile 6 months | between baseline and 6 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters probing pocket depth (PPD)
Association between PPD and GCF protein profile 12 months | between baseline and 12 months after treatment
  Change in protein profile in the gingival crevicular fluid (GCF) in relation to the clinical parameters probing pocket depth (PPD)

CONTACTS AND LOCATIONS:
Overall Officials: Lundberg, Prof., Principal Investigator — Department of Molecular Periodontology, Umeå University, Sweden
Locations (2):
- Sweden (2):
  - Specialist Clinic in Dental Care, Gävle Hospital, Public Dental Health Gävleborg AB, Region Gävleborg, Gävle, Gävleborg County
  - Specialist Clinic in Dental Care, Gävle Hospital, Public Dental Health Gävleborg, Region Gävleborg, Gävle, Gävleborg County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frencken JE, Sharma P, Stenhouse L, Green D, Laverty D, Dietrich T. Global epidemiology of dental caries and severe periodontitis - a comprehensive review. J Clin Periodontol. 2017 Mar;44 Suppl 18:S94-S105. doi: 10.1111/jcpe.12677. PMID 28266116
- [Background] Page RC. The role of inflammatory mediators in the pathogenesis of periodontal disease. J Periodontal Res. 1991 May;26(3 Pt 2):230-42. doi: 10.1111/j.1600-0765.1991.tb01649.x. PMID 1679130
- [Background] Lerner UH, Modeer T, Krekmanova L, Claesson R, Rasmussen L. Gingival crevicular fluid from patients with periodontitis contains bone resorbing activity. Eur J Oral Sci. 1998 Jun;106(3):778-87. doi: 10.1046/j.0909-8836.1998.eos106304.x. PMID 9672100
- [Background] Holmlund A, Hanstrom L, Lerner UH. Bone resorbing activity and cytokine levels in gingival crevicular fluid before and after treatment of periodontal disease. J Clin Periodontol. 2004 Jun;31(6):475-82. doi: 10.1111/j.1600-051X.2004.00504.x. PMID 15142219
- [Background] Stadler AF, Angst PD, Arce RM, Gomes SC, Oppermann RV, Susin C. Gingival crevicular fluid levels of cytokines/chemokines in chronic periodontitis: a meta-analysis. J Clin Periodontol. 2016 Sep;43(9):727-45. doi: 10.1111/jcpe.12557. Epub 2016 Jun 23. PMID 27027257
- [Background] Danesh J, Whincup P, Walker M, Lennon L, Thomson A, Appleby P, Gallimore JR, Pepys MB. Low grade inflammation and coronary heart disease: prospective study and updated meta-analyses. BMJ. 2000 Jul 22;321(7255):199-204. doi: 10.1136/bmj.321.7255.199. PMID 10903648
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] Kolny M, Stasiowski MJ, Zuber M, Marciniak R, Chabierska E, Pluta A, Jalowiecki P, Byrczek T. Randomized, comparative study of the effectiveness of three different techniques of interscalene brachial plexus block using 0.5% ropivacaine for shoulder arthroscopy. Anaesthesiol Intensive Ther. 2017;49(1):47-52. doi: 10.5603/AIT.2017.0009. PMID 28362032
- [Background] Holmlund A, Lampa E, Lind L. Poor Response to Periodontal Treatment May Predict Future Cardiovascular Disease. J Dent Res. 2017 Jul;96(7):768-773. doi: 10.1177/0022034517701901. Epub 2017 Mar 31. PMID 28363032